CLINICAL TRIAL: NCT07184996
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Phase 3, Induction Study to Evaluate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Ulcerative Colitis.
Brief Title: An Induction Study to Investigate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: SUNSCAPE-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18325; 2025-521035-37 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Duvakitug - dose 1 (Experimental): Subcutaneous (SC) injection as per protocol
  Interventions: Drug: Duvakitug
- Duvakitug - dose 2 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Placebo (Placebo Comparator): SC injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duvakitug — Pharmaceutical form:Solution for Injection-Route of administration:SC injection
  Other Names: SAR447189
  Arms: Duvakitug - dose 1; Duvakitug - dose 2
Drug: Placebo — Pharmaceutical form:Solution for injection-Route of administration:SC injection
  Arms: Placebo

SUMMARY:
This is a multinational, multicenter, randomized, double-blind, placebo-controlled, Phase 3 induction study to evaluate the efficacy and safety of duvakitug in participants with moderately to severely active Ulcerative Colitis (UC). Study details include:

The study duration may be up to 35 weeks with:

* Screening period
* 12-week Sub-Study 1 (Single-Arm Open-Label Feeder Induction) or Sub-Study 2 (Pivotal Induction)
* 12-week Sub-Study 3 (Extended Induction for non-responders)
* 45 days follow-up visit for participants who do not enroll into the maintenance study (EFC18359)

The treatment duration will be up to 12 weeks in each sub-study. The number of scheduled on-site visits will be up to 8 for the Sub-Study 1 and Sub Study 2 or a maximum of 15 visits for participants completing extended induction.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 and ≤80 years of age at Screening. Where permitted locally, participants 16 to <18 years of age who meet the definition of Tanner Stage 5 for development
* Confirmed diagnosis of moderately to severely active UC for at least 3 months prior to Baseline
* Demonstrated inadequate response, have shown loss of response or intolerance to conventional therapies or advanced therapies

Exclusion Criteria:

* Participants with Crohn's Disease (CD), indeterminate colitis
* Current diagnosis of Ulcerative Proctitis
* Participants with surgical bowel resection within the past 3 months prior to Baseline, or a history of >3 bowel resections
* Prior or current high-grade gastrointestinal (GI) dysplasia
* Participants on treatment with but not on stable doses of conventional therapies prior to baseline
* Participants with prohibited medications or therapies prior to baseline
* Participants with previous exposure to anti-TL1A investigational therapy The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-05-09 (Estimated); Study Completion 2028-05-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical remission. | Week 12
  Clinical remission is defined as modified Mayo Score (mMS) score of 0 to 2, including SFS of 0 or 1, RBS of 0, and modified Mayo Endoscopic Score (MES) of 0 or 1 (score of 1 modified to exclude friability). mMS is a composite index designed to measure UC disease activity. The score ranges from 0 to 9 with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Proportion of participants who achieve endoscopic improvement. | Week 12
  Endoscopic improvement is defined as MES of 0 or 1 (score of 1 excludes friability). Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Proportion of participants achieving clinical response by modified Mayo Score (mMS). | Week 12
  Clinical response is defined as a decrease from baseline in the mMS of ≥2 points and at least a 30% reduction from baseline, and a decrease in RB subscore of ≥1 or an absolute RB subscore of 0 or 1. mMS is a composite index designed to measure UC disease activity. The score ranges from 0 to 9 with higher scores indicating greater disease severity.
Proportion of participants achieving histological endoscopic mucosal improvement. | Week 12
  Histological endoscopic mucosal improvement is defined as MES of 0 or 1 without the evidence of friability and Geboes Score ≤3.1. The Geboes score has 6 grades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Change from baseline in PROMIS-Fatigue Short Form 7a T-score. | Baseline, Week 12
  The PROMIS-Fatigue Short Form 7 is a tool that assessesfatigue severity and its impact on daily functioning over the past week.
Proportion of participants with symptomatic (SFS and RBS) remission | Week 12
  Symptomatic remission (SF and RB): stool-frequency sub score (SFS ) of 0 or 1, and rectal bleeding sub score (RBS) of 0.
Proportion of participants with no bowel urgency. | Week 12
  The NRS for bowel urgency is a patient-reported tool designed to measure the severity of bowel urgency-the sudden or immediate need to have a bowel movement-experienced in the past 24 hours. This tool utilizes an 11-point scale for evaluation, where 0 represents "no urgency" and 10 signifies the "worst possible urgency".
Proportion of participants reporting no nocturnal bowel movements. | Week 12
Proportion of participants with symptomatic (stool-frequency sub score [SFS] and = rectal bleeding sub score [RBS]) remission. | Week 4
  Symptomatic response is defined as ≥30% decrease from baseline in the composite clinical endpoint of the sum of SFS and RBS.
Proportion of participants who achieve endoscopic remission. | Week 12
  Endoscopic remission is defined as mMES of 0.
Proportion of participants with no abdominal pain by Numeric Rating Scale (NRS). | Week 12
  The abdominal pain NRS is a tool to rate the severity of abdominal pain over the past 24 hours using a score of 0 ("no pain") to 10 ("worst possible pain").
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score. | Baseline, Week 12
  IBDQ is a tool to the quality of life of individuals suffering from IBD. The total score ranges from 32 to 224, with higher scores correlating to a better quality of life.
Proportion of participants with UC-related hospitalization. | Baseline through Week 12
Proportion of participants achieving clinical remission and no steroid use. | Week 12
Incidence of Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Adverse Events of Special Interest (TEAESIs), Treatment-Emergent Serious Adverse Events (TESAEs), and TEAEs leading to permanent study intervention discontinuation. | Baseline through 45 days after last dose
Serum concentration of duvakitug measured over time. | Baseline through Week 12
Incidence of treatment-emergent Anti-Drug Antibodies (ADA) against duvakitug. | Baseline through Week 12

CONTACTS AND LOCATIONS:
Locations (74):
- United States (60):
  - Onyx Clinical Research - Site Number: 8400021, Peoria, Arizona
  - Del Sol Research Management, LLC - Site Number: 8400012, Tucson, Arizona
  - Preferred Research Partners - Site Number: 8400018, Little Rock, Arkansas
  - FOMAT - Unio Specialty Care Arcadia - Site Number: 8400027, Arcadia, California
  - Alliance Research Institute - Site Number: 8400008, Canoga Park, California
  - Southern California GI & Liver Centers - Site Number: 8400062, Coronado, California
  - GMC Clinical Research, LLC - Site Number: 8400113, Folsom, California
  - TLC Clinical Research Inc. - Site Number: 8400030, Los Angeles, California
  - United Medical Doctors CA - Site Number: 8400044, Murrieta, California
  - Santa Maria Gastroenterology - FOMAT Medical Research HyperCORE - Site Number: 8400025, Santa Maria, California
  - Valiance Clinical Research - Tarzana - Site Number: 8400023, Tarzana, California
  - Clinical Trials Management Services - Site Number: 8400047, Thousand Oaks, California
  - Amicis Research Center-Valencia -Site Number: 8400064, Valencia, California
  - Om Research, LLC - Victorville - Site Number: 8400022, Victorville, California
  - Peak Gastroenterology Associates - Colorado Springs - Site Number: 8400039, Colorado Springs, Colorado
  - Precision Clinical Research-Site Number: 8400059, Coral Springs, Florida
  - Sarkis Clinical Trials-Ocala - Site Number: 8400048, Gainesville, Florida
  - Clinical Research of Osceola - Site Number: 8400013, Kissimmee, Florida
  - Columbus Clinical Services LLc - Site Number: 8400038, Miami, Florida
  - Regis Clinical Research, LLC - Site Number: 8400041, Miami, Florida
  - Bio Research Partner - Site Number: 8400053, Miami, Florida
  - Correa Research Center-Site Number: 8400010, Miami, Florida
  - NMC Research LLC - Site Number: 8400033, Tampa, Florida
  - M3 Wake Research - Atlanta - Site Number: 8400028, Sandy Springs, Georgia
  - EBGS Clinical Research Center, LLC - Site Number: 8400037, Snellville, Georgia
  - GI Alliance - Glenview - Site Number: 8400068, Glenview, Illinois
  - Illinois Gastroenterology Group d/b/a GI Alliance - Gurnee - Site Number: 8400049, Gurnee, Illinois
  - Gastroenterology Health Partners, PLLC - Site Number: 8400100, New Albany, Indiana
  - GI Alliance - Baton Rouge - Site Number: 8400129, Baton Rouge, Louisiana
  - GI Alliance - Metairie - Site Number: 8400124, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Mid-Atlantic GI Research, LLC - Site Number: 8400106, Greenbelt, Maryland
  - Gastroenterology Associates of Western Michigan - Site Number: 8400060, Wyoming, Michigan
  - Gateway Gastroenterology - Site Number: 8400097, Chesterfield, Missouri
  - BVL Clinical Research - Site Number: 8400005, Liberty, Missouri
  - Premier Health Research, LLC - Site Number: 8400114, Sparta, New Jersey
  - MedTraits NY - Site Number: 8400045, Maspeth, New York
  - Manhattan Clinical Research, LLC - Site Number: 8400069, New York, New York
  - New York Gastroenterology Associates - Site Number: 8400009, New York, New York
  - OnSite Clinical Solutions - Site Number: 8400051, Charlotte, North Carolina
  - Cross Creek Medical Clinic - Site Number: 8400057, Fayetteville, North Carolina
  - Monroe Biomedical Research - Site Number: 8400046, Monroe, North Carolina
  - ClinTrial Research, LLC - Site Number: 8400043, Raleigh, North Carolina
  - Plains Medical Clinic - Site Number: 8400078, Fargo, North Dakota
  - Ohio Gastroenterology Group Inc. - Site Number: 8400006, Columbus, Ohio
  - DSI Research, LLC - Site Number: 8400115, Dayton, Ohio
  - DSI Research, LLC - Site Number: 8400105, Springboro, Ohio
  - North Shore Gastroenterology Research - Site Number: 8400130, Westlake, Ohio
  - Central Sooner Research - Site Number: 8400094, Norman, Oklahoma
  - University Gastroenterology - GI Alliance - Site Number: 8400103, Providence, Rhode Island
  - Biocentric Health Research Partner, West Columbia, South Carolina
  - Valley Institute of Research - Site Number: 8400004, Harlingen, Texas
  - Innovare Research Group - Site Number: 8400067, Lake Jackson, Texas
  - Texas Digestive Disease Consultants dba GI Alliance - Lubbock - Site Number: 8400092, Lubbock, Texas
  - Texas Digestive Disease Consultants, PLLC. dba GI Alliance - Southlake - Site Number: 8400101, Southlake, Texas
  - Texas Gastro Consultants - Site Number: 8400029, Tomball, Texas
  - Tyler Research Institute, LLC - Site Number: 8400095, Tyler, Texas
  - Blue Ridge Medical Research - Site Number: 8400020, Lynchburg, Virginia
  - Clinical Research Partners - Site Number: 8400080, Richmond, Virginia
  - The Vancouver Clinic Inc. P.S. - Site Number: 8400090, Vancouver, Washington
- Canada (3):
  - Charlton Digestive Disease Centre - Site Number : 1240009, Hamilton
  - Oakville Endoscopy Center Inc. DBA ABP Research Services Corp. - Site Number : 1240010, Oakville
  - Toronto Immune and Digestive Health Institute Inc. (TIDHI) - Site Number : 1240003, Toronto
- Japan (8):
  - Asahikawa City Hospital - Site Number : 3920011, Asahikawa
  - Kagoshima IBD Gastroenterology Clinic - Site Number : 3920049, Kagoshima
  - Ofuna Chuo Hospital - Site Number : 3920029, Kamakura
  - Kokikai Tsujinaka Hospital Kashiwanoha - Site Number : 3920031, Kashiwa
  - Aoyama Clinic, Site Number : 3920018, Kobe
  - Sapporo Tokushukai Hospital - Site Number : 3920019, Sapporo
  - Tokai University Hachioji Hospital - Site Number : 3920030, Tokyo
  - Toyama University Hospital - Site Number : 3920032, Toyama
- Wellness Clinical Research - Vega Baja - Site Number: 8400099, Vega Baja, Puerto Rico
- Serbia (2):
  - Zvezdara University Medical Center, Clinic of Internal Diseases, Clinical Department of Gastroenterology and Hepatology -Site Number : 6880001, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Clinic of Internal Medicine, Department of Gastroenterology and Hepatology -Site Number : 6880002, Belgrade

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18325 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26860&tenant=MT_SNY_9011